CLINICAL TRIAL: NCT05128422
Title: Normobaric Hyperoxia Combined With Endovascular Treatment for Acute Ischemic Stroke Patients Within 6-24 Hours of Symptom Onset
Brief Title: Normobaric Hyperoxia Combined With Endovascular Treatment for Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPENS-1A
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Endovascular Treatment; Neuroprotection
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO+EVT group (Experimental): Normobaric hyperoxia Combined with Endovascular therapy group were given 100% oxygen via a face mask initiated before vascular recanalization (10L/min for 4h) . In addition, the patient will be given endovascular therapy surgery.
  Interventions: Other: Normobaric oxygen therapy
- EVT group (No Intervention): The Endovascular therapy group were given room air. And the patient will also be given endovascular therapy surgery.

INTERVENTIONS:
Other: Normobaric oxygen therapy — it is simple to administer via oxygen storage facemask at flow rates of 10 L/min for 4 hours.This therapy should begin in the emergency room as early as possible when patients meet the inclusion criteria and are randomized to the experimental group
  Arms: NBO+EVT group

SUMMARY:
The purpose of this study is to evaluate the safety and efficiency of normobaric hyperoxia combined with endovascular treatment for acute ischemic stroke patients with stroke onset 6-24 hours.

ELIGIBILITY:
Inclusion Criteria:

* age≥18;
* Suspected lage vessel occlusion of acute anterior circulation occlusion; i.e. either the ICA or the M1/M2-segment of the MCA;
* Stroke symptom onset has been more than 6 hours but not more than 24 hours,and imaging confirmed the existenceof ischemic penumbra;
* NIHSS score≥6;
* Alberta Stroke Program Early CT score (ASPECTS) of 6-10 on non- contrast CT;
* (Level of consciousness) NIHSS score of 0 or 1
* mRS score was 0-1 before stroke;
* Informed consent obtained;

Exclusion Criteria:

* Rapid improvement in neurological status to an NIHSS < 6 or evidence of vessel recanalization prior to randomization;
* Seizures at stroke onset;
* Intracranial hemorrhage;
* Systolic pressure greater than 185 mm Hg or diastolic pressure greater than 110 mm Hg, or aggressive treatment intravenous medication)necessary to reduce blood pressure to these limits;
* Symptoms rapidly improving;
* Symptoms suggestive of subarachnoid hemorrhage, even if CT scan was normal;
* Platelet count of less than 100,000 per cubic millimeter;
* CT showed a multiple infarction (low density area greater than 1/3 cerebral hemisphere);
* severe hepatic or renal dysfunction;
* active and chronic obstructive pulmonary disease or acute respiratory distress syndrome;
* >3 L/min oxygen required to maintain peripheral arterial oxygen saturation (SaO2)#95% as per current stroke management guidelines;
* medically unstable;
* inability to obtain informed consent;
* Life expectancy<90 days;
* Pregnant or breast-feeding women;
* Unwilling to be followed up or poor compliance for treatment;
* Patients being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial;
* Evidence of intracranial tumor;
* Baseline blood glucose of < 50 mg/dL (2.78 mmol) or > 400 mg/dL (22.20 mmol);
* Patients with upper gastrointestinal bleeding or nausea and vomiting who cannot use oxygen masks;
* Other circumstances requiring emergency oxygen inhalation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Early neurologic improvement (ENI) at 24 hours | 24 ± 12 hours
  ENI was defined as percent change NIHSS≥30%; Percent change NIHSS was defined as [(admission NIHSS score-24-hour NIHSS score)x100/admission NIHSS score];

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale(NIHSS) Score | 4 hours ± 15 minutes, 24 ± 12 hours; 7 ± 2 days after randomization
  the NIHSS is a stroke severity score that is composed of 11 items; range from 0 to 42, higher values indicate more severe deficits
modified Rankin Scale score (mRS) | 90 ± 14 days after randomization
  secondary clinical efficacy endpoint;the mRs is an ordinal disability score of 7 categories (0 = no symptoms to 5 = severe disability, and 6 = death)
Change in National Institutes of Health Stroke Scale (NIHSS) score from baseline to 24 hours | 24 ± 12 hours after randomization
  secondary clinical efficacy endpoint;the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits)
Barthel Index (BI) | 90 ± 14 days after randomization
  secondary clinical efficacy endpoint;the BI is an ordinal disability score of 10 categories(range from 0 to 100, higher values indicate better prognosis);
Revascularization on 24-hour follow-up imaging | 24 ± 12 hours hours after randomization
  secondary imaging efficacy endpoint;Successful recanalization was defined as mTICI 2b or 3
Early neurologic deterioration | 24 ± 12 hours after randomization
  NIHSS score increased by more than 4 points);the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits);clinical safety endpoint;
Symptomatic Intracerebral Hemorrhage | 24± 12 hours hours after randomization
  imaging safety endpoints;Deterioration in NIHSS score of ≥4 points within 24 hours;per ECASS III definition and per Heidelberg bleeding classification
Mortality | 90 ± 14 days after randomization
  clinical safety endpoint;
Stroke recurrence | 90 ± 14 days，180 ± 30 days after randomization
  clinical safety endpoint;
The 5-level EuroQol five dimensions questionnaire（EQ-5D-5L）score | 90 ± 14 days after randomization
  secondary clinical efficacy endpoint, Quality of Life score; The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Delta NIHSS | 24 ± 12 hours after randomization
  Delta NIHSS was defined (admission NIHSS score-24-hour NIHSS score).
Percent change NIHSS | 24 ± 12 hours after randomization
  Percent change NIHSS was defined as [(admission NIHSS score-24-hour NIHSS score)x100/admission NIHSS score]
Cerebral infarct volume | 36 ± 12 hours after randomization
  Infarct volume is evaluated mainly through brain MRI(DWI) or CT

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, China